CLINICAL TRIAL: NCT05818540
Title: Randomized Controlled Trial to Compare Effectiveness of DreamPort-Eclipse to a Traditional Nasal Mask
Brief Title: Sleep Apnea Study in Adults Using DreamPort-Eclipse and a Traditional Nasal Mask
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bleep, LLC (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSL-SNAP-003; 1R44HL158286-01A1 (NIH)
Record Dates: First submitted 2023-04-04; First posted 2023-04-19 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Masking Description: Data collected will be deidentified upon collection - surveys and assessment forms will be labelled with a numerical identifier.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Eclipse novel mask (Experimental): Human subjects will use the Eclipse CPAP interface for 60 days for a total of 6 hours per night.
  Interventions: Device: Eclipse novel CPAP mask
- Traditional CPAP mask (Active Comparator): Human subjects will use the ResMed P-10 CPAP interface for 60 days for a total of 6 hours per night.
  Interventions: Device: ResMed P-10 mask

INTERVENTIONS:
Device: Eclipse novel CPAP mask — Participants will wear the mask for 6 hours a night for 60 days.
  Arms: Eclipse novel mask
Device: ResMed P-10 mask — Participants will wear the mask for 6 hours a night for 60 days.
  Arms: Traditional CPAP mask

SUMMARY:
The Randomized Controlled Trial of Bleep DreamPort-Eclipse Study is a two-arm, randomized, prospective, non-blinded study to assess the effectiveness of the novel CPAP human interface design to improve leak, AHI, and pressure compared to a traditional nasal mask.

ELIGIBILITY:
Inclusion Criteria:

• Male or female ≥18 years old who are impacted by obstructive sleep apnea and currently are familiar with a CPAP device

Exclusion Criteria:

* Any medical or behavioral conditions that would compromise subject safety
* Under the age of 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Heatherington, Principal Investigator — Bleep, LLC
Locations (1):
- Sleep Centers of Middle Tennessee, Murfreesboro, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected through surveys will be available upon request to the principal investigator. Data requested will be de-identified. Only de-identified data will be made available. Only survey responses and the investigators' observational notes, also deidentified, will be shared. No PHI will be shared. Aggregated participant demographic data will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available 4 years after the study completion.
Access Criteria: Requests will be made in writing, to the PI, at stuart@bleepsleep.com. Requests should include the reason for the request, how the data is intended to be used, and additional information may be requested. Data will be shared with credentialed, licensed, or otherwise verifiable researchers/investigators for research purposes only.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Newly diagnosed OSA patients, were recruited from SCMT centers.
Period: Overall Study
Arm/Group | Eclipse Novel Mask | Traditional CPAP Mask
Started | 74 (Participated, started in trial) | 99 (Participated, started in trial)
Completed | 30 | 54
Not Completed | 44 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eclipse Novel Mask | Traditional CPAP Mask | Total
Number analyzed (Participants) | 30 | 54 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 53 | 83
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.2) | 58.5 (9.5) | 47.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 24 | 38
  Male | 16 | 30 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Completed participants: White | 19 | 43 | 62
  Completed participants: Black | 10 | 7 | 17
  Completed participants: Hispanic | 1 | 4 | 5
  Completed participants: Asian | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index (AHI)
Description: AHI recorded from the software built-in algorithm. The Apnea-Hypopnea Index or Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. The apneas (pauses in breathing) must last for at least 10 seconds and be associated with a decrease in blood oxygenation.
Time Frame: 60 days
Population: Participants who used the Eclipse or P10 mask over a period of 60 days and completed the trial.
Measure: Mean (Standard Deviation); unit: events/h
Groups:
- Eclipse Novel Mask: Human subjects used the Eclipse CPAP interface for 60 days for a total of 6 hours per night.
Arm/Group | Eclipse Novel Mask | Traditional CPAP Mask
Number analyzed (Participants) | 30 | 54
events/h | 2.7 (3.3) | 2.5 (4.7)

2. Primary Outcome: Leak
Description: Data were captured from the device in L/min at 60 days. Leak is how much flow in L exits the mask while the patient wears it each min. It is recorded through proprietary algorithm undisclosed to the public by the device
Time Frame: 60 days
Population: Participants who used the Eclipse or P10 mask over a period of 60 days and completed the trial.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Eclipse Novel Mask | Traditional CPAP Mask
Number analyzed (Participants) | 30 | 54
L/min | 3.66 (5.38) | 3.01 (3.36)

3. Primary Outcome: CPAP Device Pressure (P95)
Description: Therapeutic positive pressure (in cmH2O) that the device administer for 95% of the night. It is recorded through proprietary algorithm undisclosed to the public by the device.
Time Frame: 60 days
Population: Participants who used the Eclipse or P10 mask over a period of 60 days and completed the trial.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Eclipse Novel Mask | Traditional CPAP Mask
Number analyzed (Participants) | 30 | 54
cmH2O | 8.93 (1.01) | 8.62 (1.46)

4. Secondary Outcome: Participant Satisfaction With the Mask Choice
Description: A 16-item patient survey was administered to the participants in each arm at the end of the study. Patients had to answer according to a Likert scale (1: worst, 5:best). This reflects the average of all the answered items. For example, question number one had an average score of 4.48 for the eclipse mask arm and 4.12 for the standard mask arm, question number 2 had an average score of 4.40 for the eclipse mask arm and 4.42 for the standard mask arm, etc. Since all questions reflect participant satisfaction, they were averaged to provide an overall score.
Time Frame: 60 days
Population: Participants who used the Eclipse or P10 mask over a period of 60 days and completed the trial.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Eclipse Novel Mask | Traditional CPAP Mask
Number analyzed (Participants) | 30 | 54
score | 4.3 (0.4) | 4.1 (0.4)

5. Secondary Outcome: Percentage of Participants Who Could Tolerate the Mask Well (Mask Tolerability)
Description: We estimated the mask tolerability as follows (as a percentage): 100*(participants who completed the trial) / [(participants who completed the trial) + (participants who discontinued the trial due to a desire to switch masks or poor mask compliance)].
Time Frame: 60 days
Population: Participants who used the Eclipse or P10 mask over a period of 60 days and completed the trial.
Measure: Number; unit: % of enrolled participants
Arm/Group | Eclipse Novel Mask | Traditional CPAP Mask
Number analyzed (Participants) | 30 | 54
% of enrolled participants | 41 | 55

ADVERSE EVENTS:
Time Frame: 6 months
Description: There were no adverse events reported.
Arm/Group | Eclipse Novel Mask | Traditional CPAP Mask
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/54
Other Adverse Events (participants affected / at risk) | 0/30 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT05818540/Prot_SAP_000.pdf